CLINICAL TRIAL: NCT02203123
Title: Ratio of Inferior Vena Cava and Aorta Diameter in Dehydrated Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Hee Lee, Assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ultrasound_01
Record Dates: First submitted 2014-06-17; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration | interventions — Ultrasonography; Saline Solution

ARMS (1):
- Ultrasound, inferior vena cava, aorta, normal saline (Other)
  Interventions: Device: Ultrasound; Drug: normal saline

INTERVENTIONS:
Device: Ultrasound
Drug: normal saline

SUMMARY:
* There is no definite tool for measurement of dehydration in children
* Subjective clinical dehydration scale is considered as valuable scoring system, but it cannot be reliable among clinicians sometimes.
* Some authors found Inferior vena cava/Aorta ratio can be a objective marker for dehydration
* However, there is no evidence of correlation between clinical dehydration scale and inferior vena cava/aorta ratio
* We will observe correlation between clinical dehydration scale and inferior vena cava/aorta ratio and change of the ratio according to hydration with intravenous normal saline infusion.

ELIGIBILITY:
Inclusion Criteria:

* All children with dehydration who visit emergency department

Exclusion Criteria:

* congenital heart disease
* bronchopulmonary dysplasia
* renal disease
* liver disease

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 226 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
diameter of inferior vena cava and aorta | up to 2 hours
  we will measure the diameter of inferior vena cava and aorta using ultrasound during every 10 ml/kg infusion of intravenous normal saline

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hee Lee, Professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Gumi-dong, Seongnam-si, Gyeonggi-do, South Korea